CLINICAL TRIAL: NCT05902858
Title: Efferct of Standard Laryngoscopy Versus Video-laryngoscop on First-attempt Success in Difficult Airways Undergoing ProVu TM Video Stylet Guided Intubationa (PROVU)
Brief Title: Effect of Standard Laryngoscopy Versus Video-laryngoscopy
Acronym: PROVU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Flexicare Medical Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASO.RianGen.22.03
Record Dates: First submitted 2023-01-23; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-01

CONDITIONS: Difficult Intubation
Keywords: PROVU; Videolaryngoscopy; Laryngoscopy
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Intervention Model Description: open-label, randomized, 3-parallel arm, monocentric trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Conventional intubation with hyperangulated videolaryngoscope
  Interventions: Device: Conventional intubation with hyperangulated videolaryngoscope
- Provu TM video stylet + hyperangulated videolaryngoscope (Experimental): Intubation ProVu TM video stylet combined with hyperangulated videolaryngoscope
  Interventions: Device: Intubation with ProVu TM video stylet combined with hyperangulated videolaryngoscope
- Provu TM video stylet + Macintosh laryngoscope (Experimental): Intubation ProVu TM video stylet combined with standard Macintosh laryngoscope
  Interventions: Device: Intubation with ProVu TM video stylet combined with standard Macintosh laryngoscope

INTERVENTIONS:
Device: Conventional intubation with hyperangulated videolaryngoscope — After the induction of general anesthesia, the patient will undergo conventional intubation with hyperangulated videolaryngoscope
  Arms: Control Group
Device: Intubation with ProVu TM video stylet combined with hyperangulated videolaryngoscope — After the induction of general anesthesia, the patient will undergo intubation with ProVu TM video stylet combined with hyperangulated videolaryngoscope
  Arms: Provu TM video stylet + hyperangulated videolaryngoscope
Device: Intubation with ProVu TM video stylet combined with standard Macintosh laryngoscope — After the induction of general anesthesia, the patient will undergo intubation with ProVu TM video stylet combined with standard Macintosh laryngoscope
  Arms: Provu TM video stylet + Macintosh laryngoscope

SUMMARY:
The aim of this open-label, randomized, 3-parallel arm trial is to compare success of intubation rate at first try between three groups that will be intubated:

1. Conventional intubation with hyperangulated videolaryngoscope (control group),
2. Intubation ProVu TM video stylet combined with hyperangulated videolaryngoscope,
3. Intubation ProVu TM video stylet combined with standard Macintosh laryngoscope.

DETAILED DESCRIPTION:
Critical anesthetic incidents in the operating room are often related to airway management. Difficult airway management is defined as the clinical situation in which an anesthesiologist with conventional training has difficulty with upper airway face mask ventilation, difficulty with tracheal intubation, or both. Airway management has undergone a major transformation since the development of hyper-angle videolaryngoscopy (VL). Recently, the ProVuTM video stylet (Flexicare Medical Ltd, Mountain Ash, UK), which combines visualization technology with a tube guidance system, has been proposed as a new device for endotracheal intubation in participants with difficult airway management.

The investigators hypothesized that the ProVuTM video stylet combined with videolaryngoscopy or standard laryngoscopy may improve the success rate of intubation on the first attempt compared with using a videolaryngoscope alone in patientes with predicted difficult intubation. In fact, using ProVuTM the position of the video stylet tip can be adjusted continuously during the tracheal intubation maneuver.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective surgery requiring oral tracheal intubation;
* ≥18 years of age;
* simplified Arné score ≥11;
* Written informed consent will be obtained from every participant.

Exclusion Criteria:

* ≤18 years of age
* interincisor distance at maximal mouth opening ≤2 cm;
* planned awake fiberoptic intubation because patients are patients considered to be high-risk for difficult intubation or difficult mask ventilation (e.g. with neck tumours, complete cervical arthrodesis; neck circumference >50 cm);
* patients at risk of gastric aspiration
* planned nasal intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Success rate on first intubation attemps | During the procedure
  The first-attempt intubation success is defined as tracheal tube placement with a single maneuver after insertion of the tube in the mouth. Reinsertion of the tube in the mouth counts as an additional attempt.

SECONDARY OUTCOMES:
Time of intubation | During the procedure
  Time from insertion of the laryngoscope beyond the dental rhyme to cuffed tube
Time of laryngoscopy | During the procedure
  Time from insertion of the laryngoscope beyond the dental rhyme to the insertion of the tube beyond the dental rhyme
Number of intubation attempts | During the procedure
  Times of reinsertion of the tube beyond the dental rhyme
Complications | During the procedure
  Evaluation of the type and rate of complications, including desaturation < 90%, esophageal intubation, tooth breakage and bleeding from the oropharyngeal mucosa
Use of "jaw trust" or "BURP" | During the procedure
  Need to perform adjuvant maneuvers (jaw trust or BURP), measured with yes/no
Need of another anesthesiologist intervention | During the procedure
  Required intervention of another anesthesiologist, measured with yes/no, after 3 failed intubation attempt or after request of the first anesthesiologist
Needs to change the path of the intubation strategy | During the procedure
  Needs to change intubation strategy, measured with yes/no, includes use of fiberoptic intubation, change of videolaryngoscope or postpone intervention
Learning curve analysis of intubation rate success | Through study completion, an average of 1 year
  Improvement of intubation rate success
Learning curve analysis of time of procedure | Through study completion, an average of 1 year
  Improvement of time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Leo, Physician, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrison SL, Ahmad I, Elwen F, Curtis A, Dua G, Surda P, Johnstone C. Awake tracheal intubation with the ProVu video stylet: a case series. Anaesth Rep. 2021 Mar 29;9(1):e12102. doi: 10.1002/anr3.12102. eCollection 2021 Jan-Jun. PMID 33817645